CLINICAL TRIAL: NCT02727114
Title: Echographic Imaging Research to the Anatomical and Physiological Characteristics of the Skin in Children and Adolescents
Brief Title: Echographic Measurement of Skin Thickness in Children
Acronym: PIDIC-1
Status: Completed | Type: Observational
Sponsor: Novosanis NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015_NOV_VX_003
Record Dates: First submitted 2016-03-23; First posted 2016-04-04 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Skin Thickness
Keywords: skin thickness; high-frequency ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- participants aged 8 weeks to 3 years: Echographic measurement of skin thickness at the proximal forearm, the deltoid region and medial thigh (till age of 2 years) in participants aged 8 weeks to 3 years.
  aimed number: 32 boys & 32 girls / maximum number: 50 boys & 50 girls
  Interventions: Other: Echographic measurement of skin thickness
- participants aged 3 to 6 years: Echographic measurement of skin thickness at the proximal forearm and the deltoid region in participants aged 3 to 6 years.
  aimed number: 32 boys & 32 girls / maximum number: 50 boys & 50 girls
  Interventions: Other: Echographic measurement of skin thickness
- participants aged 6 to 12 years: Echographic measurement of skin thickness at the proximal forearm and the deltoid region in participants aged 6 to 12 years.
  aimed number: 32 boys & 32 girls / maximum number: 50 boys & 50 girls
  Interventions: Other: Echographic measurement of skin thickness
- participants aged 12 to 18 years: Echographic measurement of skin thickness at the proximal forearm and the deltoid region in participants aged 12 to 18 years.
  aimed number: 32 boys & 32 girls / maximum number: 50 boys & 50 girls
  Interventions: Other: Echographic measurement of skin thickness

INTERVENTIONS:
Other: Echographic measurement of skin thickness — (Epi)Dermal thickness at the proximal forearm, the deltoid region and medial site of the thigh (till 2 years) will be measured using imaging technology, more specifically high-frequency ultrasound (20-70 MHz) in B-mode (VEVO 2100® & VEVO 3100®, Visual Sonics). This non-invasive measuring technique has already been proven to be accurate.
  The echographic measurement will be performed on the left and right deltoid and medial thigh region, and on two sides of the proximal forearm. Both the dorsal part and the volar/palmar part of the proximal forearm will be investigated. Ultrasound will be executed using gel (Aquasonic®) to optimize imaging.

SUMMARY:
To optimize a medical device for intradermal injection, knowledge concerning the thickness of epidermis and dermis at the proximal forearm is required. Since scientific knowledge is lacking, the investigators will examine the skin thickness (epidermis and dermis) of children (aged 8 weeks to 18 years) using imaging technology (High Frequency Ultrasound). The investigators hypothesize that they are able to correlate the thickness of the (epi)dermis to a specific combination of parameters age, gender, and BMI.

Based on these results, the investigators can define which needle type and length is needed to correctly perform injections into the dermal layer

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Age: 8 weeks to 18 years
* Dutch-speaking
* Caucasian

Exclusion Criteria:

* Using ointment, crème, gels or oral medication based on corticoids
* Suffering from skin diseases (psoriasis, burning wounds)
* Pregnancy or lactating

Ages: 8 Weeks to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be recruited in the vicinity of the university and its university hospital of Antwerp. Through primary and secundary school in Antwerp, children will be recruited after approval of their parents and via some Child and Family (Dutch: Kind&Gezin) facilities children aged 8 weeks to 3 years will recruited.
  All recruitement will be done from October 2015 until November 15th 2015.
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
skin thickness (in millimeters) of the proximal dorsal forearm (both left and right) | 5-10 minutes
skin thickness (in millimeters) of the proximal ventral forearm (both left and right) | 5-10 minutes
skin thickness (in millimeters) of the deltoid region (both left and right) | 5-10 minutes
skin thickness (in millimeters) of the medial thigh region (both left and right) | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Vankerckhoven, PhD, Principal Investigator — CEO
Locations (3):
- Belgium (3):
  - University of Antwerp, Wilrijk, Antwerp
  - Child & Family (Dutch: Kind&Gezin) Antwerp, Antwerp
  - primary and secundary schools in Antwerp, Belgium, Antwerp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Mulder TJS, Van Nuffel D, Demolder M, De Meyer G, Moens S, Beyers KCL, Vankerckhoven VVJ, Van Damme P, Theeten H. Skin thickness measurements for optimal intradermal injections in children. Vaccine. 2020 Jan 22;38(4):763-768. doi: 10.1016/j.vaccine.2019.11.002. Epub 2019 Nov 22. PMID 31767463